CLINICAL TRIAL: NCT03614481
Title: Clinical and Genetic Analyzes of Age-related Macular Degeneration
Acronym: COLDMLA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: COLLECTION DMLA; 2013-A00110-45 (Other: ID-RCB)
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — salivary swabs, venous sampling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AMD patient: During the AMD consultation, patients have their imaging exams including OCT, retinophotography, and fluorescein angiography.
  After the interview with the doctor on pathology diagnosis and follow-up, they will meet the clinical research associate nurse to complete the questionnaire and perform anthropometric measurements (weight, height, abdominal perimeter measurement and blood pressure measurement). Patients recruited at Créteil will benefit from a venous blood sample (20 mL) in 2 EDTA tubes for DNA extraction after light reading and signature of consent. For patients recruited from other ophthalmic centers, the Clinical Research Associate will perform salivary sampling for DNA extraction after light reading and signature of consent.
  Interventions: Genetic: Sampling
- control without AMD: 898/5000 Given the observation of a mutation in an unaffected control individual, it is not excluded that this individual may be suffering from AMD at a later age. The observation of the mutation could thus be considered as a pre-clinical test. None of the teams were able to obtain a control population of the same age and sex ratio, which could have benefited from fluorescein angiography or at least a fundus examination, to ensure the absence of warning signs of AMD. This requires cooperation from healthy elderly volunteers not only for blood sampling but also for pupillary dilatation.
  The controls may be the accompanying persons or spouses of AMD patients. It may also be people seen in general consultation without maculopathy or retinopathy with an age greater than 55 years.
  Interventions: Genetic: Sampling

INTERVENTIONS:
Genetic: Sampling — Sampling

SUMMARY:
The purpose of this collection is to search for susceptibility genes for age-related macular degeneration (AMD) alone or in combination with environmental factors and to look for genes that modulate the AMD phenotype (particularly the response to treatment).

ELIGIBILITY:
Inclusion Criteria:

* Age> 55 years
* Diagnosis of exudative or atrophic AMD in at least one eye
* Patient informed of the objectives of the study and having freely signed the informed consent letter
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Other retinal or choroidal lesion in the studied eye
* History of severe systemic disease that could potentially hinder patient adherence to the study protocol: mental disorder, cancer, recent stroke or heart failure less than 3 months old.
* Known allergy to fluorescein, indocyanine green, iodine or ranibizumab

Min Age: 55 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Diagnosis of exudative or atrophic AMD
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2005-11 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Genotypic factors | 6 months
  Identification of genotypic factors associated with good or poor response to treatment in precisely phenotyped AMD patients.

SECONDARY OUTCOMES:
Predictive markers | 6 months
  Look for predictive markers of cure response among polymorphisms that are susceptibility factors for AMD
Vascular Endothelial Growth Factor | 6 months
  Look for predictors of treatment response among polymorphisms of other genes: Vascular Endothelial Growth Factor, Vascular Endothelial Growth Factor Receptor
Environmental factors | 6 months
  Look for predictive markers of treatment response among environmental factors
Predictive treatment response score | 6 months
  Create a predictive treatment response score that combines factors independently associated with the response to treatment in multivariate analysis
Circulating biological factors | 6 months
  Identification of circulating biological factors such as circulating fatty acids at risk of AMD or modulating the response to treatment.

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Hôpital Pellegrin, Bordeaux
  - CHI Créteil, Créteil
  - Hôpital général de Dijon, Dijon
  - Hôpital des Quinze-Vingts, Paris
  - Centre ophtalmologique d'imagerie et de laser, Paris

IPD SHARING:
Plan to Share IPD: No